CLINICAL TRIAL: NCT00410462
Title: Randomized Phase II Study of Brostallicin (PNU-166196A) Versus Doxorubicin as First Line Chemotherapy in Patients With Advanced or Metastatic Soft Tissue Sarcoma
Brief Title: Brostallicin or Doxorubicin as First-Line Therapy in Treating Patients With Relapsed, Refractory, or Metastatic Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-62061; EORTC-62061; EUDRACT-2006-001861-40; NERVIANO-BRTA-0100-015
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2010-07

CONDITIONS: Ovarian Cancer; Sarcoma; Small Intestine Cancer
Keywords: recurrent adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; adult liposarcoma; adult fibrosarcoma; adult malignant fibrous histiocytoma; adult leiomyosarcoma; adult rhabdomyosarcoma; adult alveolar soft-part sarcoma; adult malignant mesenchymoma; adult angiosarcoma; adult epithelioid sarcoma; adult neurofibrosarcoma; adult synovial sarcoma; recurrent uterine sarcoma; stage IV uterine sarcoma; ovarian sarcoma; small intestine leiomyosarcoma; recurrent small intestine cancer
MeSH Terms: conditions — Ovarian Neoplasms; Sarcoma; Liposarcoma; Fibrosarcoma; Histiocytoma, Malignant Fibrous; Leiomyosarcoma; Rhabdomyosarcoma; Sarcoma, Alveolar Soft Part; Malignant mesenchymal tumor; Hemangiosarcoma; Neurofibrosarcoma; Sarcoma, Synovial | interventions — brostallicin; Doxorubicin

INTERVENTIONS:
Drug: brostallicin
Drug: doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as brostallicin and doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This randomized phase II trial is studying the side effects and how well brostallicin or doxorubicin works as first-line therapy in treating patients with relapsed, refractory, or metastatic soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the activity and safety of brostallicin vs doxorubicin hydrochloride as first-line therapy in patients with relapsed, refractory, or metastatic soft tissue sarcoma.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating and age(younger than 60 years vs 60 years and over). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive brostallicin IV over 10 minutes on day 1.
* Arm II: Patients receive doxorubicin hydrochloride IV over 10 minutes on day 1. In both arms, treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 30 days and then every 12 weeks thereafter.

PROJECTED ACCRUAL: A total of 108 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed high- or intermediate-grade malignant soft tissue sarcoma* of 1 of the following cellular types:

  * Adipocytic (e.g., liposarcoma dedifferentiated, myxoid/round cell, pleomorphic, mixed-type, not otherwise specified)
  * Fibroblastic (e.g., adult fibrosarcoma, myxofibrosarcoma, or sclerosing epithelioid fibrosarcoma)
  * So-called fibrohistiocytic (e.g., pleomorphic malignant fibrous histiocytoma [MFH], giant cell MFH, or inflammatory MFH)
  * Leiomyosarcoma
  * Malignant glomus tumors
  * Skeletal muscle (e.g., rhabdomyosarcoma, alveolar, or pleomorphic)
  * Vascular (e.g., epithelioid hemangioendothelioma or angiosarcoma)
  * Uncertain differentiation (e.g., synovial, epithelioid, alveolar soft part, clear cell, desmoplastic small round cell, extra-renal rhabdoid, malignant mesenchymoma, perivascular epithelioid cell tumor [PEComa], or intimal sarcoma)
  * Malignant peripheral nerve sheath tumors
  * Malignant solitary fibrous tumors
  * Undifferentiated soft tissue sarcomas not otherwise specified
  * Other types of sarcoma if approved by the study coordinator NOTE: *Includes malignant tumors of non-organ origin and skin and uterine leiomyosarcoma
* The following tumor types are excluded:

  * Embryonal rhabdomyosarcoma
  * Chondrosarcoma
  * Osteosarcoma
  * Ewing tumors/primitive neuroectodermal tumor (PNET)
  * Gastrointestinal stromal tumors
  * Dermatofibrosarcoma protuberans
  * Inflammatory myofibroblastic sarcoma
  * Neuroblastoma
  * Malignant mesothelioma
  * Mixed mesodermal tumors of the uterus
* Relapsed, refractory, and/or metastatic disease incurable by surgery or radiotherapy
* Measurable disease
* Must have formalin fixed paraffin-embedded tumor blocks and representative hematoxylin/eosin slides available for histological central review
* No symptomatic or known CNS metastases

PATIENT CHARACTERISTICS:

* At least 60 years of age OR ≥ 18 years of age if patient is not suitable for intensive combination chemotherapy treatments
* WHO performance status 0-1
* Absolute neutrophil count > 2,000/mm³
* Platelet count > 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Creatinine clearance ≥ 60 mL/min
* No serious cardiac illness within the past 6 months, including, but not limited to the following:

  * History of documented congestive heart failure
  * High-risk uncontrolled arrhythmias
  * Angina pectoris requiring antianginal medication
  * Clinically significant valvular heart disease
  * Evidence of transmural infarction on ECG
  * Poorly-controlled hypertension (e.g., systolic blood pressure [BP] > 180 mm Hg or diastolic BP > 100 mm Hg)
* Normal 12-lead ECG
* LVEF normal by MUGA or echocardiogram
* No other malignancy within the past 3 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast
* No other serious and/or unstable medical condition, illness, or lab abnormality that would preclude study participation
* No psychiatric illness or familial, social, or geographical condition that would preclude study compliance
* No active uncontrolled infection
* No known AIDS positivity
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy regimen for advanced or metastatic disease (neoadjuvant and adjuvant therapy allowed)
* No concurrent sargramostim (GM-CSF) except in cases of febrile neutropenia
* No other concurrent anticancer therapy or investigational agents, including any of the following:

  * Chemotherapy
  * Biological response modifiers
  * Hormone therapy
  * Immunotherapy
* No other concurrent clinical treatment trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2006-10; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Six-month progression-free survival, in terms of complete response, partial response, or no change

SECONDARY OUTCOMES:
Overall progression-free survival
Objective tumor response
Safety (CTCAE v 3.0)
Duration of response
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Hans Gelderblom, MD, PhD, Study Chair — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Result] Gelderblom H, Blay JY, Seddon BM, Leahy M, Ray-Coquard I, Sleijfer S, Kerst JM, Rutkowski P, Bauer S, Ouali M, Marreaud S, van der Straaten RJ, Guchelaar HJ, Weitman SD, Hogendoorn PC, Hohenberger P. Brostallicin versus doxorubicin as first-line chemotherapy in patients with advanced or metastatic soft tissue sarcoma: an European Organisation for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group randomised phase II and pharmacogenetic study. Eur J Cancer. 2014 Jan;50(2):388-96. doi: 10.1016/j.ejca.2013.10.002. Epub 2013 Nov 8. PMID 24215845